CLINICAL TRIAL: NCT01996358
Title: Comparing Intubating Conditions Using Succinylcholine or Rocuronium/Sugammadex for Rigid Bronchoscopy: a Randomized Study
Brief Title: Comparing Intubating Conditions Using Succinylcholine or Rocuronium for Rigid Bronchoscopy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Grietje Beck, Professor Dr. med, Dr. Horst Schmidt Klinik GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK004
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Intubating Conditions; Postoperative Myalgia; Patient Satisfaction
Keywords: Succinylcholine; Rocuronium; Rigid Bronchoscopy
MeSH Terms: conditions — Patient Satisfaction | interventions — Succinylcholine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Succinylcholine (Active Comparator): Succinylcholine 0,5mg/kg as muscle relaxant during induction of anaesthesia for rigid bronchoscopy
  Interventions: Drug: Succinylcholine
- Rocuronium 0,3 (Active Comparator): Rocuronium 0,3 mg/kg during induction of anaesthesia for rigid bronchoscopy. At the end of procedure 2mg/kg sugammadex for reversal of neuromuscular block are applied.
  Interventions: Drug: Rocuronium 0,3
- Rocuronium 0,6 (Active Comparator): Rocuronium 0,6 mg/kg during induction of anaesthesia for rigid bronchoscopy. At the end of procedure 2mg/kg sugammadex for reversal of neuromuscular block are applied.
  Interventions: Drug: Rocuronium 0,6

INTERVENTIONS:
Drug: Succinylcholine — Anaesthesia is induced and maintained with propofol (1-2 mg/kg) and remifentanil (0,5 µg/kg). The study arm is immobilized and after cleaning the skin a dual electrode for peripheral nerve stimulation is placed over the ulnar nerve near the wrist. Neuromuscular monitoring is performed with accelerometry. After induction of anaesthesia the patient receives muscle relaxant according to the study group.
  Arms: Succinylcholine
Drug: Rocuronium 0,3 — General anaesthesia is induced and maintained with propofol (1-2mg/kg) and remifentanil (0,5µg/kg). The study arm is immobilized and after cleaning the skin a dual electrode for peripheral nerve stimulation is placed over the ulnar nerve near the wrist. Neuromuscular monitoring is performed with accelerometry. The Patient receives the muscle relaxant according to the study group.
  Arms: Rocuronium 0,3
Drug: Rocuronium 0,6 — General anaesthesia is induced and maintained with propofol (1-2mg/kg) and remifentanil (0,5µg/kg). The study arm is immobilized and after cleaning the skin a dual electrode for peripheral nerve stimulation is placed over the ulnar nerve near the wrist. Neuromuscular monitoring is performed with accelerometry. The Patient receives the muscle relaxant according to the study group.
  Arms: Rocuronium 0,6

SUMMARY:
Succinylcholine is commonly used for neuromuscular relaxation for short procedures such as rigid bronchoscopy. A more modern alternative is the application aof rocuronium, reversed by sugammadex. The investigators compare the intubating conditions, incidence of postoperative myalgia (POM) as well as patient satisfaction for these two muscle relaxants.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yr
* scheduled for elective rigid bronchoscopy

Exclusion Criteria:

* known neuromuscular disease
* significant hepatic or renal dysfunction
* family history of malignant hyperthermia
* known allergy to one of the drugs used in this protocol
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Intubating Condition | after induction of general anaesthesia (after 3-5 minutes)
  The intubating conditions will be measured using the scoring system proposed for Good Clinical Research Practice using the following variables: conditions of inserting the rigid bronchoscope, vocal cord position and coughing

SECONDARY OUTCOMES:
Postoperative Myalgia | 72 hours after intervention
  The severity of POM is measured by using a four-point-scale:
  0. no myalgia
  1. minor pain limited to one area of the body
  2. muscle pain or stiffness noticed spontaneously by the patient, which may have required analgesic therapy
  3. generalized, severe or incapacitating discomfort

OTHER OUTCOMES:
Patient satisfaction | 72 hours after intervention
  measurement on a numeric ten point scale

CONTACTS AND LOCATIONS:
Overall Officials: Grietje Beck, Prof, Study Chair — Dr. Horst Schmidt Klinik
Locations (1):
- Dr. Horst Schmidt Klinik, Wiesbaden, Hesse, Germany